CLINICAL TRIAL: NCT02086435
Title: A Randomized Controlled Trial on Intracorporeal Versus Extracorporeal Morcellation With Endobag Extraction in Patients Undergoing Laparoscopic Myomectomy: Clinical Efficacy and Safety Outcomes
Brief Title: Intracorporeal Versus Extracorporeal Morcellation: Clinical Efficacy and Safety Outcomes
Acronym: IEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SafeMorcellation
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Uterine Myoma
Keywords: Myomectomy; Laparoscopic myomectomy; Morcellation; Risk of dissemination; Uterine Sarcoma; Parasitic myoma
MeSH Terms: conditions — Myofibroma | interventions — Morcellation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal morcellation (Experimental): Extracorporeal morcellation in which patients are treated with "protected" removal by endobag and extracorporeal myoma morcellation with cold scissors and scalpel blade or with power morcellator used inside the bag itself
  Interventions: Procedure: Extracorporeal morcellation
- Intracorporeal morcellation (Active Comparator): Intracorporeal morcellation patients treated with standard intracorporeal morcellation, using reusable electronic device
  Interventions: Procedure: Intracorporeal morcellation

INTERVENTIONS:
Procedure: Extracorporeal morcellation — patients treated with "protected" removal by endobag and extracorporeal myoma morcellation with cold scissors and scalpel blade or with power morcellator used inside the bag itself
  Other Names: protected morcellation; morcellation in endobag
  Arms: Extracorporeal morcellation
Procedure: Intracorporeal morcellation — patients treated with standard intracorporeal morcellation, using reusable electronic device
  Other Names: Power morcellation; Standard intracorporeal morcellation
  Arms: Intracorporeal morcellation

SUMMARY:
The aim of this study protocol will be to compare the technique of intracorporeal morcellation using reusable electronic device (standard technique) with a technique of removal "protected" by endobag and extracorporeal myoma morcellation with cold scissors and scalpel blade or with power morcellator used inside the bag itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopy for uterine myomas with international guidelines surgical indications
* Presence of at least one uterine myoma larger than 4 cm
* Aged between 18 and 40 years

Exclusion Criteria:

* Presence of uterine neoformations suspicious for malignancy
* Medical major disorders associated
* Acute or chronic psychiatric disorders
* Ascertained Premenstrual syndrome
* Use of drugs that can affect cognitive ability or state of consciousness and alertness during the last six months prior to enrollment
* Presence of calcified fibroids ultrasound examination
* Presence of adnexal lesions
* Detection of a pattern of endometrial hyperplasia with atypia determined in the course endometrial biopsy performed for abnormal uterine bleeding
* Abnormal PAP test
* Positive Pregnancy Test
* Previous use of laparoscopic surgery increased

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Operative time | The day of surgery
  calculated from the time, after secured hemostasis of the uterine breach, in which the myoma is clamped and subjected to intracorporeal or added in endobag for extracorporeal morcellation to the moment when the 'last fragment of myoma will be considered removed from the surgical field

SECONDARY OUTCOMES:
Total operative time | The day of surgery
  from skin incision to skin closure
Handling of morcellation | The day of surgery
  expressed on the VAS scale where 1 means very bad handling and 10 excellent handling
Blood loss | 2 hours after the end of surgery
  Blood loss will be calculated by the difference of Hb level 2 hours after surgery and the morning of the surgery
Postoperative hospital stay | The day of patient discharge, average 4 day after surgery
Postoperative pain | The day of patient discharge, average 4 day after surgery
  measured on the VAS scale where 1 stands for a little pain and 10 for intense pain
Rate of complications | The day of patient discharge, average 4 day after surgery
  need of transfusion or laparotomic conversion

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy

REFERENCES:
- [Derived] Venturella R, Rocca ML, Lico D, La Ferrera N, Cirillo R, Gizzo S, Morelli M, Zupi E, Zullo F. In-bag manual versus uncontained power morcellation for laparoscopic myomectomy: randomized controlled trial. Fertil Steril. 2016 May;105(5):1369-1376. doi: 10.1016/j.fertnstert.2015.12.133. Epub 2016 Jan 19. PMID 26801067